CLINICAL TRIAL: NCT04852432
Title: Evaluation of the Efficacy of Oxygen Therapy and Clinical Feasibility of High Flow Nasal Cannula During Moderate and Deep Sedation in Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H2103-095-1205
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Pediatric Sedation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Nasal prong is applied, but sedation is performed without oxygen administration.
- Low flow group (Experimental): Oxygen administration by nasal cannula
  Interventions: Device: nasal prong
- High flow group (Experimental): Oxygen is administered at a rate of 2L/kg/min using an Optiflow device
  Interventions: Device: high flow nasal cannula

INTERVENTIONS:
Device: high flow nasal cannula — The heated air is administered at a rate of 2L/kg/min using an Optiflow device (Fisher and Paykel Healthcare, Auckland, New Zealand). Inhalation oxygen concentration starts with 50%.
  Arms: High flow group
Device: nasal prong — Oxygen is administered via nasal prong
  Arms: Low flow group

SUMMARY:
The investigators evaluate the efficacy and safety of routine administration of oxygen during moderate or deep sedation in pediatric patients. In addition, in terms of efficacy and safety, oxygen administration via nasal prong and high flow nasal cannula will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Children under the age of 18 who undergo moderate-deep sedation

Exclusion Criteria:

* Respiratory failure patients
* Increased intracranial pressure
* Recent massive nasal bleeding
* History of airway surgery
* Complete nasal obstruction
* Pulmonary hypertension
* Skull base fracture

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 258 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Desaturation (≤95%) | through study completion, average 30 minutes
  Occurrence of desaturation (pulse oximeter ≤95%)

SECONDARY OUTCOMES:
Desaturation (≤90%) | through study completion, average 30 minutes
  Occurrence of desaturation (pulse oximeter ≤90%)
CO2 value | through study completion, average 30 minutes
  percutaneous CO2 (maximum, minimum, mean values)
Minimum saturation during sedation | through study completion, average 30 minutes
Complications | through study completion, average 30 minutes
  Any complications during sedation

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Ko HJ, Park JB, Ji SH, Kim JT. Oxygen Supplementation in Pediatric Sedation: Prospective, Multicenter, Randomized Controlled Trial. Anesthesiology. 2025 Jul 1;143(1):132-141. doi: 10.1097/ALN.0000000000005500. Epub 2025 Apr 11. PMID 40215365